CLINICAL TRIAL: NCT01250197
Title: A Double-masked, Crossover Study Assessing the Ocular and Systemic Safety and Systemic Absorption of Two Formulations of 0.5% AR-12286 Ophthalmic Solution in Normal Volunteers
Brief Title: Formulation Comparison in Normal Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aerie Pharmaceuticals (Industry)
Responsible Party: Thomas van Haarlem, M.D., Aerie
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AR-12286-CS101
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2010-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Normal Volunteers
Keywords: Normal Volunteers
MeSH Terms: interventions — AR-12286

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Formulation A (Experimental): AR-12286 Ophthalmic Solution Formulation A
  Interventions: Drug: AR-12286
- Formulation B (Experimental): AR-12286 Ophthalmic Solution Formulation B
  Interventions: Drug: AR-12286

INTERVENTIONS:
Drug: AR-12286 — Ophthalmic Solution

SUMMARY:
This is a double-masked, single-center, crossover study in which normal volunteers will be randomized to receive one of two formulations of 0.5% AR-12286 Ophthalmic Solution for 8 days. Subjects will undergo a minimum 7-day washout, and then receive the alternate treatment for 8 days.

DETAILED DESCRIPTION:
Not desired.

ELIGIBILITY:
Inclusion Criteria:

* Normal volunteers

Exclusion Criteria:

* Active ophthalmic or systemic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2010-11; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Ocular safety | 3 weeks
  The primary safety endpoints will be visual acuity, objective biomicroscopic and ophthalmoscopic examination, and subjective comfort as measured by adverse events in response to subject symptom queries.

CONTACTS AND LOCATIONS:
Overall Officials: Tom van Haarlem, MD, Study Director — Aerie Pharmaceuticals, Inc.
Locations (1):
- Celerion, Phoenix, Arizona, United States